CLINICAL TRIAL: NCT00060801
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of 24 Weeks of Oral Treatment With BIIL 284 BS in Adult (75 mg, 150 mg) and Pediatric (75 mg) Cystic Fibrosis Patients
Brief Title: Efficacy and Safety of 24 Weeks of Oral Treatment With BIIL 284 BS in Adult and Pediatric Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Purpose: Treatment
Other Study IDs: BI 543.45
Record Dates: First submitted 2003-05-13; First posted 2003-05-14 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; BIIL 284; Boehringer Ingelheim
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Drug: BIIL 283 BS (Amelubent)

SUMMARY:
The purpose of this study is to determine the effect of 24 weeks of treatment with BIIL 284 BS compared with placebo on pulmonary function and incidence of pulmonary exacerbation in adult and pediatric cystic fibrosis patients.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female patients >= 6 years pediatric 6-17 years inclusive; adult >= 18 years)
* Body weight >= 20 kg (determined at Visit 1)
* Confirmed diagnosis of CF
* Able to perform acceptable spirometric maneuvers, according to American Thoracic Society standards .
* FEV1 25-85% predicted
* Clinically stable
* The patient or the patient's legally acceptable representative must be able to give informed consent.
* The patient must be able to swallow the BIIL 284 BS tablets whole.
* Patients taking a chronic medication must be willing to continue this therapy for the entire duration of the study.

EXCLUSION CRITERIA:

* Patients with a significant history of allergy/hypersensitivity (including medication allergy) which is deemed relevant to the trial as judged by the Investigator. "Relevance" in this context refers to any increased risk of hypersensitivity reaction to trial medication; there are no specific issues of concern currently identified with respect to use of BIIL 284 BS in allergic patients per se.
* Patients who have participated in another study with an Investigational drug within one month or 6 half-lives (whichever is greater) preceding the screening visit.
* Patients with known relevant substance abuse, including alcohol or drug abuse.
* Female patients who are pregnant or lactating, including females who have a positive serum pregnancy test at screening (pregnancy tests will be performed for all females of child bearing potential).
* Female patients of child bearing potential who are not using a medically approved form of contraception.
* Patients who are unable to comply with food requirements prior to dosing.
* Patients with documented persistent colonization with Burkholderia cepacia.
* Patients chronically using oral corticosteroids or high-dose ibuprofen.
* Patients with hemoglobin < 9.0 g/dL; platelets < 100x10 to the 9th power/L; SGOT (ALT) or SGPT (AST) > 2.5 times the upper limit of normal; creatinine > 1.5 times upper limit normal.
* Clinically significant disease or medical condition other than Cystic Fibrosis or Cystic Fibrosis-related conditions that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420
Dates: Start 2003-05; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in post-bronchodilator forced expiratory volume in one second (FEV1) (percent predicted) | 28 weeks
Proportion of patients with at least one pulmonary exacerbation during the treatment period as per definition of Fuchs et al | 28 weeks

SECONDARY OUTCOMES:
Change from baseline in post-bronchodilator forced vital capacity (FVC) percent predicted | 28 weeks
Change from baseline in post-bronchodilator mean forced expiratory flow during the middle half of the FVC (FEF25-75% ) percent predicted | 28 weeks
Change from baseline in post-bronchodilator maximal expiratory flow when 50% of FVC remains in lung (MEF50% )percent predicted | 28 weeks
Change from baseline in post-bronchodilator maximal expiratory flow when 25% of FVC remains in lung (MEF25%) percent predicted | 28 weeks
Change from baseline in post-bronchodilator inspiratory capacity (IC) | 28 weeks
Change from baseline in post-bronchodilator slow vital capacity (SVC) | 28 weeks
Change from baseline in pre-bronchodilator FEV1% predicted | week 12, 24 and 28
Change from baseline in pre-bronchodilator FVC % predicted | week 12, 24 and 28
Change from baseline in pre-bronchodilator FEF25-75% % predicted | week 12, 24 and 28
Change from baseline in pre-bronchodilator MEF50% % predicted | week 12, 24 and 28
Change from baseline in pre-bronchodilator MEF25%% predicted | week 12, 24 and 28
Proportion of patients with at least one pulmonary exacerbation during the treatment period as described in Rosenfeld et al. | 28 weeks
Time to first pulmonary exacerbation | 28 weeks
Number of pulmonary exacerbations during the treatment period | 28 weeks
Proportion of patients with at least 1 hospitalisation for a pulmonary exacerbation during the treatment period | 28 weeks
Time to first hospitalisation for a pulmonary exacerbation | 28 weeks
Number of hospitalisations for a pulmonary exacerbation | 28 weeks
Number of days in hospital for a pulmonary exacerbation | 28 weeks
Proportion of patients with at least one pulmonary exacerbation requiring i.v. antibiotics during the treatment period | 28 weeks
Time to first course of i.v. antibiotics for a pulmonary exacerbation | 28 weeks
Number of pulmonary exacerbations requiring i.v. antibiotics during the treatment period | 28 weeks
Number of days of i.v. antibiotic use for pulmonary exacerbations during the treatment period | 28 weeks
Change from baseline in weight | 28 weeks
Change from baseline in height (in pediatrics) | 28 weeks
Change from baseline in weight for age percentiles | 28 weeks
Change from baseline in weight for age percentiles (in pediatrics) | 28 weeks
Change from baseline in weight expressed as % ideal body weight (IBW) | 28 weeks
Change from baseline in body mass index | 28 weeks
Change from baseline in BMI for age percentiles | 28 weeks
Change from baseline in blood levels of cytokines, chemokines and other inflammatory mediators | 28 weeks
Change in patient's health status as reported by patient | 28 weeks
Change in patient's health status as reported by physician | 28 weeks

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Children's Hospital & Health Center, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - The Nemours Children's Clinic, Orlando, Florida
  - Pediatric Pulmonary Associates, PA, St. Petersburg, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Riley Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University-St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Albany Medical College, Albany, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - MCP Hospital, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Children's Memorial Center of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Wisconsin Hospitals & Clinics, Madison, Wisconsin